CLINICAL TRIAL: NCT00820404
Title: Ascending Single Dose Study of the Safety, Tolerability, and Pharmacokinetics of BLI-489 Administered Intravenously to Healthy Subjects
Brief Title: Study Evaluating Single Doses of BLI-489 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3219K1-1000
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — BLI-489

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): BLI-489
  Interventions: Drug: BLI-489
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BLI-489
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety, and tolerability of single doses of BLI-489 administered intravenously in healthy subjects, and also how the drug is absorbed and eliminated.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women of nonchildbearing potential, 18 to 50 years of age inclusive at screening.
2. Body mass index (BMI) in the range of 18 to 32 kg/m2 and body weight greater than or equal to 50 kg.
3. Healthy as determined by the investigator on the basis of the screening evaluations.
4. Nonsmoker of smoker of fewer than 10 cigarettes per day as determined by history.

Exclusion Criteria:

1. Presence of history of any disorder that may prevent the successful completion of the study.
2. History of drug abuse within 1 year.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety as measured by the number of adverse events and serious adverse events. Tolerability will be assessed based upon the occurrence of dose limiting toxicities. | 15 days

SECONDARY OUTCOMES:
Pharmacokinetics as evaluated by drug concentrations in the blood and urine. | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Philadelphia, Pennsylvania, United States